CLINICAL TRIAL: NCT00187278
Title: Biventricular Pacing for Atrioventricular Block in Left Ventricular Dysfunction to Prevent Cardiac Desynchronization
Brief Title: Biopace Study: Biventricular Pacing for Atrioventricular Block to Prevent Cardiac Desynchronization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR03006HF
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Atrioventricular Block; Ventricular Dysfunction
Keywords: Standard pacing indication
MeSH Terms: conditions — Atrioventricular Block; Ventricular Dysfunction | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RV Pacing (Active Comparator): Standard Pacemaker implant
  Interventions: Device: RV Pacing
- Biventricular Pacing (Experimental): Biventricular Pacemaker implant
  Interventions: Device: Biventricular Pacing

INTERVENTIONS:
Device: Biventricular Pacing — Biventricular Pacemaker implant
  Arms: Biventricular Pacing
Device: RV Pacing — Standard Pacemaker implant
  Arms: RV Pacing

SUMMARY:
The primary purpose of the study is to evaluate if patients with a standard indication for permanent ventricular pacing, left ventricular ejection fraction without limit, or any QRS duration will profit from the prevention of ventricular desynchronisation.

DETAILED DESCRIPTION:
The study will be performed as a controlled, single-blind, international, multicenter, prospective, randomized, parallel group design.

In order to pragmatically examine the effectiveness of biventricular pacing in patients with an indication for ventricular pacing, the study group with biventricular pacing is compared to a control group with standard pacemakers which only allow univentricular (right ventricular) stimulation, as it has been the standard outside of clinical studies until so far.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of an indication for ventricular pacing according to the actual guidelines for the implantation of cardiac pacemakers and a need for frequent (or even permanent) ventricular pacing for:

   1. Permanent 3rd degree atrioventricular (AV)-block or
   2. Intermittent 3rd degree AV-block in combination with 1st degree AV-block with a pQ-interval ≥ 220 ms or
   3. 2nd degree AV-block type Mobitz II in combination with 1st degree AV-block with a pQ-interval ≥ 220 ms or
   4. 2nd degree AV-block type Mobitz I (if indicated) in combination with 1st degree AV-block with a pQ-interval ≥ 220 ms or
   5. 1st degree AV-block with a pQ-interval ≥ 220 ms and indication for ventricular pacing (includes indication for ventricular pacing based on long HV interval measured during invasive electrophysiological testing) or
   6. Sick-sinus-syndrome with symptomatic sinus bradycardia or sinus arrest as primary indication for device implantation in combination with long 1st degree AV-block with a pQ-interval ≥ 220 ms or
   7. Chronic (permanent) atrial fibrillation (flutter or tachycardia) with a spontaneous heart (ventricular) rate at rest ≤ 60/min or
   8. Chronic (permanent) atrial fibrillation (flutter or tachycardia) with a spontaneous heart (ventricular) rate at rest ≤ 75/min, if initiation or increase of pharmacological treatment with a relevant heart rate lowering effect (negative chronotropic effect) is planned for the time after pacemaker implantation (i.e. ß-blockers for heart failure and rate control)
   9. Patients scheduled for AV node ablation
2. Any QRS duration and morphology
3. Left ventricular ejection fraction (LVEF) without limit as measured by echocardiography (in at least one plane, either 4- or 2-chamber or apical long axis view)
4. Signed written informed consent of the patient or a first-degree relative for study participation after informing the patient/relative about the risks and the aim of the study
5. Willingness and ability to comply with the prescribed follow-up tests and schedule of evaluations.
6. Absence of an implanted ventricular pacing device (patients with atrial pacemakers and new need for ventricular pacing may be included)

Exclusion Criteria:

1. Implanted Cardioverter Defibrillator or consideration for implantation of an ICD due to arrhythmia indication. However, ICD implant for primary prevention of sudden cardiac death in patients with LVEF ≤ 35 % (in accordance with the actual guidelines for the implantation of arrhythmia devices[LVEF < 30%] and in accordance with the results of the SCD-Heft study [LVEF < 35%) will be allowed.
2. Implanted ventricular pacing device
3. Status 1 for cardiac transplantation and likelihood to receive transplantation within 2 years (these patients would not be expected to fulfill the follow-up requirements as outlined in this protocol)
4. Evidence of acute left ventricular dysfunction and high probability for its reversibility (e.g. acute myocarditis, tachycardiomyopathy)
5. Implanted prosthetic tricuspid valve
6. Severe musculoskeletal disorder(s)
7. Age below 18 years
8. Current or planned pregnancy in the next 6 months
9. Current or recent (within the past 30 days) participation in any other clinical investigation
10. Life expectancy of less than 6 months
11. Patient's inability to independently comprehend and complete the Quality of Life (QoL) questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1833 (Actual)
Dates: Start 2003-05; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Funck, MD, Principal Investigator — Klinikum Bad Hersfeld, Germany; Jean-Jacques Blanc, Prof., Study Chair — Hôpital Cavale Blanche, Brest, France
Locations (1):
- Klinikum der Philipps-Universität Marburg, Marburg, Germany

REFERENCES:
- [Background] Funck RC, Blanc JJ, Mueller HH, Schade-Brittinger C, Bailleul C, Maisch B; BioPace Study Group. Biventricular stimulation to prevent cardiac desynchronization: rationale, design, and endpoints of the 'Biventricular Pacing for Atrioventricular Block to Prevent Cardiac Desynchronization (BioPace)' study. Europace. 2006 Aug;8(8):629-35. doi: 10.1093/europace/eul075. PMID 16864616
- [Background] Funck RC, Mueller HH, Lunati M, Piorkowski C, De Roy L, Paul V, Wittenberg M, Wuensch D, Blanc JJ; BioPace study group. Characteristics of a large sample of candidates for permanent ventricular pacing included in the Biventricular Pacing for Atrio-ventricular Block to Prevent Cardiac Desynchronization Study (BioPace). Europace. 2014 Mar;16(3):354-62. doi: 10.1093/europace/eut343. Epub 2013 Nov 7. PMID 24200715
- [Derived] Funck RC, Muller HH, Lunati M, De Roy L, Klein N, Meisel E, Milasinovic G, Carlson MD, Wittenberg M, Hindricks G, Blanc JJ. Biventricular vs. right ventricular pacing devices in patients anticipated to require frequent ventricular pacing (BioPace). Europace. 2025 Mar 5;27(3):euaf029. doi: 10.1093/europace/euaf029. PMID 40105785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between May 2003 and September 2007.
Pre-assignment Details: 1834 patients have been scheduled for randomization, while 1833 have been randomized to RV Pacing or Biventricular group.
  One patient could not be randomized due to organizational reasons.
Period: Overall Study
Arm/Group | RV Pacing | Biventricular Pacing
Started | 918 | 915
Completed | 908 | 902
Not Completed | 10 | 13
Not completed — Protocol Violation | 10 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RV Pacing | Biventricular Pacing | Total
Number analyzed (Participants) | 908 | 902 | 1810
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (9.0) | 73.8 (9.0) | 73.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 296 | 278 | 574
  Male | 612 | 624 | 1236
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (4.7) | 27.4 (4.3) | 27.4 (4.5)
Ventricular pacing at 1 month [Mean (Inter-Quartile Range); unit: %] | 86.4 [48 to 88] | 90.2 [67 to 93] | 88.3 [56 to 91]
Underlying cardiac diseases [Number; unit: participants]
  All | 572 | 571 | 1143
  Ischaemic heart disease | 274 | 274 | 548
  Hypertensive heart disease | 281 | 262 | 543
  Dlated cardiomyopathy | 43 | 51 | 94
  Valvulopathy | 170 | 165 | 335
  Prior MI | 162 | 141 | 308
Cardiovascular risk factor [Number; unit: participants] — Some participants experienced more than one cardiovascular risk factor.
  participants
    Hypertension | 696 | 666 | 1362
    Diabetes mellitus | 255 | 251 | 506
Left ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: %] | 55.5 (12.4) | 55.3 (12.1) | 55.4 (12.2)
Left Ventricular Ejection Fraction (LVEF) range [Number; unit: participants]
  LVEF ≤ 35% | 74 | 78 | 152
  35% < LVEF ≤ 50% | 221 | 198 | 419
  LVEF > 50% | 613 | 626 | 1239
QRS duration [Mean (Standard Deviation); unit: ms] | 118.8 (30.3) | 118.1 (30.8) | 118.4 (30.5)
QRS range [Number; unit: participants]
  QRS ≤ 120ms | 571 | 571 | 1142
  120ms < QRS ≤ 150ms | 190 | 176 | 366
  QRS > 150ms | 147 | 155 | 302
Atrial arrhythmias [Number; unit: participants]
  Atrial arrhythmias | 225 | 225 | 450
  None | 683 | 677 | 1360
Left bundle branch block (LBBB) [Number; unit: participants]
  LBBB | 166 | 150 | 316
  None | 742 | 752 | 1494
Scheduled for ICD [Number; unit: participants]
  Scheduled for ICD | 22 | 26 | 48
  Not scheduled for ICD | 886 | 976 | 1762
Indications for device implantation [Number; unit: participants]
  Persistent bradycardia | 538 | 540 | 1078
  Intermittent bradycardia | 368 | 362 | 730
  Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Total Mortality
Description: Number of deaths observed
Time Frame: Study duration (5.7 years mean follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 908 | 902
Participants | 307 | 305
Statistical Analysis 1: Comparison: RV Pacing vs Biventricular Pacing; Test type: Superiority or Other; p = 0.3492, Regression, Cox — adjusted p; Hazard Ratio (HR) = 0.926, 95% CI 2-sided [0.789 to 1.0088]

2. Primary Outcome: Death or Heart Failure Hospitalization
Description: Number of subjects who experienced death or hospitalization where heart failure is a primary cause of hospitalization
Time Frame: Study duration (5.7 years mean follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 908 | 902
Participants | 346 | 363
Statistical Analysis 1: Comparison: RV Pacing vs Biventricular Pacing; Test type: Superiority or Other; p = 0.0882, Regression, Cox — adjusted p; Hazard Ratio (HR) = 0.878, 95% CI 2-sided [0.756 to 1.020]

3. Secondary Outcome: Death Due to Cardiovascular Causes
Description: Number of subjects who died due to cardiovascular causes, as classified by the independent Event Adjudication Committee (IEAC)
Time Frame: Study duration (5.7 years mean follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 908 | 902
Participants | 106 | 107
Statistical Analysis 1: Comparison: RV Pacing vs Biventricular Pacing; Test type: Superiority or Other; p = 0.8215, Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.74 to 1.27]

4. Secondary Outcome: Functional Capacity as Measured by the Distance Covered in the 6-minute Walk Test
Time Frame: 12 months post-implant
Population: This analysis includes all enrolled patients who completed the 6-minute walk test both at the baseline and 12-month visits. Due to that reason, the overall number of participants analyzed is different from the participant module.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 672 | 675
meters | 371.3 (128.8) | 371.2 (129.1)

5. Secondary Outcome: Health Related Quality of Life Measured by the Minnesota Living With Heart Failure Questionnaire©
Description: Minnesota Living with Heart Failure (MLWHF) questionnaire score at 12 months
  MLWHF score: the total scale is from 0 to 105, with higher scores indicating worse health status.
Time Frame: 12 months post-implant
Population: This analysis includes all enrolled patients who completed the Minnesota Living With Heart Failure questionnaire both at the baseline and 12-month visits. Due to that reason, the overall number of participants analyzed is different from the participant module.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 724 | 715
score on a scale | 16.0 (15.4) | 15.3 (15.5)

6. Secondary Outcome: Incidence of Hospitalizations for Deterioration of Heart Failure
Time Frame: Study duration (5.7 years mean follow-up)
Measure: Number; unit: hospitalization per patient year
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 899 | 888
hospitalization per patient year | 0.043 | 0.037

7. Secondary Outcome: Incidence of Hospitalizations for Cardiovascular Events
Time Frame: Study duration (5.7 years mean follow-up)
Measure: Number; unit: hospitalizations per patient year
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 899 | 888
hospitalizations per patient year | 0.162 | 0.161

8. Secondary Outcome: Incidence of Hospitalizations for Any Reason
Time Frame: Study duration (5.7 years mean follow-up)
Measure: Number; unit: Hospitalization per patient year
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 899 | 888
Hospitalization per patient year | 0.392 | 0.432

9. Secondary Outcome: Cardiac Structure and Function
Time Frame: 12 & 24 months
Population: Data related to cardiac structure and function can not be presented as the data was not collected and analysis provided by the core lab.
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Successful Implantation of the Left Ventricular Lead
Time Frame: Implantation
Population: There was an attempt of left ventricular lead implantation only for subjects from Biventricular Pacing group.
Measure: Number; unit: participants
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 0 | 883
participants |  | 760

11. Secondary Outcome: Chronic Atrial Fibrillation (Defined as Presence of Atrial Fibrillation in Two Subsequent ECG´s/Visits)
Description: Chronic atrial fibrillation is defined as presence of atrial fibrillation in two subsequent ECG´s/visits.
Time Frame: Study duration (5.7 years mean follow-up)
Measure: Number; unit: participants
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 908 | 902
participants | 91 | 76

12. Secondary Outcome: Functional Capacity as Measured by the Distance Covered in the 6-minute Walk Test
Time Frame: 24 months post-implant
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 614 | 592
meters | 369.3 (127.2) | 376.5 (132.0)

13. Secondary Outcome: Health Related Quality of Life Measured by the Minnesota Living With Heart Failure Questionnaire©
Description: Minnesota Living with Heart Failure (MLWHF) questionnaire score at 24 months.
  MLWHF score: the total scale is from 0 to 105, with higher scores indicating worse health status.
Time Frame: 24 months post-implant
Population: This analysis includes all enrolled patients who completed the Minnesota Living With Heart Failure questionnaire both at the baseline and 24-month visits. Due to that reason, the overall number of participants analyzed is different from the participant module.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 662 | 675
score on a scale | 17.5 (17.6) | 17.3 (16.6)

14. Secondary Outcome: Duration of Hospitalizations for Deterioration of Heart Failure
Time Frame: Study Duration (5.7 years mean follow-up)
Measure: Number; unit: days per patient year
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 899 | 888
days per patient year | 0.40 | 0.39

15. Secondary Outcome: Duration of Hospitalizations for Cardiovascular Events
Time Frame: Study Duration (5.7 years mean follow-up)
Measure: Number; unit: Days per patient year
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 899 | 888
Days per patient year | 1.52 | 1.50

16. Secondary Outcome: Duration of Hospitalizations for Any Reason
Time Frame: Study duration (5.7 years mean follow-up)
Measure: Number; unit: days per patient year
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 899 | 888
days per patient year | 3.72 | 4.14

17. Secondary Outcome: Adverse Events Related to Left Ventricular Lead
Description: Only serious adverse events related to the left ventricular lead are included.
Time Frame: Study Duration (5.7 years mean follow-up)
Measure: Number; unit: participants
Arm/Group | RV Pacing | Biventricular Pacing
Number analyzed (Participants) | 908 | 902
participants | 1 | 38

ADVERSE EVENTS:
Time Frame: Study duration (5.7 years mean follow-up)
Description: The sponsor assessed all events except the death cases without further information, duplicate events and uncomplicated device replacement due to end of life. 5628 events were reviewed and assessed by the sponsor. Subjects may experience more than one adverse event.
Arm/Group | RV Pacing | Biventricular Pacing
All-Cause Mortality (participants affected / at risk) | 307/908 | 305/902
Serious Adverse Events (participants affected / at risk) | 641/908 | 698/902
Other Adverse Events (participants affected / at risk) | 451/908 | 507/902
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RV Pacing (N=908) | Biventricular Pacing (N=902)
Anemia (Blood and lymphatic system disorders) | 14 (19) | 14 (16)
Epistaxis (Blood and lymphatic system disorders) | 3 (3) | 2 (2) — device pocket revision, lead dysfunction.
Haemoptysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hematochezia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypercalcemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thromboemboli (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
AV Fistula (Cardiac disorders) | 1 (1) | 3 (5)
Acute Coronary Syndrome (Cardiac disorders) | 5 (7) | 1 (1)
Angina (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 48 (56) | 54 (75)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (3)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Chest Pain (Cardiac disorders) | 50 (68) | 48 (63)
Dyspnea (Cardiac disorders) | 46 (71) | 60 (74)
Endocarditis (Cardiac disorders) | 2 (2) | 5 (7)
Exacerbation of heart failure (Cardiac disorders) | 132 (179) | 103 (144)
Hypertension (Cardiac disorders) | 13 (16) | 18 (20)
Hypertrophic obstructive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 5 (5) | 5 (5)
Mitral Regurgitation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 29 (34) | 26 (26)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3)
Rise in threshold and exit block (Cardiac disorders) | 12 (12) | 22 (24)
Shortness of Breath (Cardiac disorders) | 4 (4) | 3 (3)
Valve damage (Cardiac disorders) | 26 (36) | 18 (19)
Lowry Wood Syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 4 (4)
Diabetes (Endocrine disorders) | 10 (13) | 12 (12)
Glycemia (Endocrine disorders) | 0 (0) | 2 (2)
Hyperglycemia (Endocrine disorders) | 2 (2) | 4 (4)
Hypoglycemia (Endocrine disorders) | 3 (5) | 5 (6)
Cataract (Eye disorders) | 2 (3) | 1 (1)
Galucoma (Eye disorders) | 1 (1) | 1 (1)
Macular Degeneration (Eye disorders) | 0 (0) | 1 (1)
Cholangitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 4 (6) | 3 (4)
Ulcer (Gastrointestinal disorders) | 2 (2) | 4 (6)
Antral gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastroenteritis (Gastrointestinal disorders) | 4 (4) | 2 (2)
Hernia (Gastrointestinal disorders) | 16 (16) | 8 (8)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 15 (17) | 16 (18)
Drug Toxicity (General disorders) | 1 (1) | 0 (0)
Dysphagia (General disorders) | 0 (0) | 1 (1)
Dysphonia (General disorders) | 0 (0) | 1 (1)
Esophagitis (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 11 (11) | 12 (13)
Hospitalization for non-cardiac diseases (General disorders) | 74 (86) | 87 (110)
Hydrocephalus (General disorders) | 0 (0) | 1 (1)
Influenza (General disorders) | 5 (5) | 1 (1)
Lyme Disease (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 47 (57) | 55 (65)
Shingles (General disorders) | 0 (0) | 1 (1)
Stenosis (General disorders) | 22 (22) | 17 (20)
Syncope (General disorders) | 22 (25) | 17 (18)
Weakness (General disorders) | 6 (6) | 4 (5)
Worsening of General Patient's Condition (General disorders) | 39 (47) | 59 (65)
Cirrhosis (Hepatobiliary disorders) | 1 (1) | 3 (3)
Gallbladder disease (Hepatobiliary disorders) | 2 (2) | 2 (2)
Gallstones (Hepatobiliary disorders) | 1 (1) | 8 (11)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy (Immune system disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 58 (76) | 87 (118)
Sepsis (Infections and infestations) | 6 (6) | 7 (10)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Abdominal adhesions post surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental injury (Injury, poisoning and procedural complications) | 2 (2) | 8 (8)
Acute hemorrhage/bleeding (Injury, poisoning and procedural complications) | 26 (27) | 35 (39)
Air emboli (Injury, poisoning and procedural complications) | 9 (11) | 10 (10)
Amputation (Injury, poisoning and procedural complications) | 5 (7) | 8 (9)
Cardiac or venous perforation (Injury, poisoning and procedural complications) | 6 (6) | 9 (9)
Cardiac/coronary sinus dissection (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Coronary sinus or cardiac vein thrombosis (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Erosion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excessive bleeding (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Extracardiac stimulation (phrenic nerve, diaphragm, chest wall) (Injury, poisoning and procedural complications) | 1 (1) | 12 (12)
Fall (Injury, poisoning and procedural complications) | 33 (34) | 39 (42)
Hematoma/seroma formation (Injury, poisoning and procedural complications) | 14 (22) | 19 (19)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication Error (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pericardial effusion (Injury, poisoning and procedural complications) | 1 (1) | 8 (10)
Pericarditis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pleural Effusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bone fracture (Musculoskeletal and connective tissue disorders) | 24 (28) | 32 (37)
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Adenomatous polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (26) | 32 (36)
Local tissue reaction; formation of fibrotic tissue; cyst formation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (20) | 16 (16)
Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33 (40) | 35 (48)
Concussion (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Nervous system disorders) | 4 (4) | 4 (4)
Dimentia (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 4 (4) | 4 (5)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 4 (4) | 2 (2)
Radicular syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Sleep Apnea (Nervous system disorders) | 1 (1) | 2 (2)
Inappropriate mode switch (Product Issues) | 0 (0) | 1 (1)
Inappropriate shocks (Product Issues) | 1 (1) | 0 (0)
Lead Fracture (Product Issues) | 2 (2) | 1 (1)
Lead migration, dislodgment or poor lead placement (Product Issues) | 31 (37) | 36 (39)
Loss of Capture (Product Issues) | 3 (3) | 6 (6)
Mechanical malfunction of the pacing lead (Product Issues) | 2 (3) | 1 (1)
Oversensing (Product Issues) | 3 (4) | 2 (2)
Pacemaker Mediated Tachycardia (Product Issues) | 2 (2) | 0 (0)
Pacing Lead Impedance Out of Range (Product Issues) | 3 (3) | 3 (4)
Pulse Generator Reset (Product Issues) | 0 (0) | 1 (1)
Undersensing (Product Issues) | 2 (2) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 0 (0) | 1 (1)
Cardiac or venous perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Kidney Stones (Renal and urinary disorders) | 1 (2) | 0 (0)
Kidney disease (Renal and urinary disorders) | 8 (8) | 7 (9)
Macrohematuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Nephrocalcinosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Disease (Renal and urinary disorders) | 11 (12) | 20 (20)
Renal failure (Renal and urinary disorders) | 16 (17) | 21 (22)
Ureteral Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Track Disease (Renal and urinary disorders) | 6 (6) | 5 (8)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 (18) | 17 (21)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 52 (58) | 36 (41)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 16 (24)
Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 11 (15)
Abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Colposcopy (Surgical and medical procedures) | 0 (0) | 2 (2)
Coronary artery bypass surgery (Surgical and medical procedures) | 1 (1) | 3 (3)
Endoscopic Retrograde Cholangiopancreatography (Surgical and medical procedures) | 1 (1) | 0 (0)
Iron Infusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Percutaneous Coronary Intervention (Surgical and medical procedures) | 27 (32) | 19 (27)
Planned Lead Revision (Surgical and medical procedures) | 1 (1) | 0 (0)
Planned Pulse Generator Replacement (Surgical and medical procedures) | 191 (201) | 306 (335)
Pulse Generator Pocket Revision (Surgical and medical procedures) | 1 (1) | 2 (3)
Surgery (Surgical and medical procedures) | 77 (89) | 80 (101)
Aneurysm (Vascular disorders) | 7 (10) | 4 (4)
Cerebrovascular Accident (Vascular disorders) | 5 (5) | 9 (10)
Coronary artery disease (Vascular disorders) | 5 (5) | 4 (5)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Fluid accumulation (Vascular disorders) | 26 (32) | 35 (39)
Lim Ischemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 3 (3) | 2 (2)
Peripheral artery disease (Vascular disorders) | 0 (0) | 2 (2)
Stroke (Vascular disorders) | 21 (27) | 26 (29)
Transient Ischemic Attack (Vascular disorders) | 16 (18) | 26 (28)
Venous occlusion (Vascular disorders) | 2 (3) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RV Pacing (N=908) | Biventricular Pacing (N=902)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 1 (2) | 3 (3)
Hematochezia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypereosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thromboemboli (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 96 (119) | 107 (135)
Arteritis (Cardiac disorders) | 0 (0) | 1 (1)
Bigeminy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 24 (29) | 31 (43)
Dyspnea (Cardiac disorders) | 38 (47) | 47 (55)
Exacerbation of heart failure (Cardiac disorders) | 23 (24) | 23 (23)
Heart block (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 8 (9) | 13 (15)
Hypotension (Cardiac disorders) | 7 (9) | 8 (8)
Mitral Regurgitation (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 9 (9) | 4 (4)
Palpitations (Cardiac disorders) | 7 (8) | 4 (6)
Percutaneous Coronary Intervention (Cardiac disorders) | 0 (0) | 1 (1)
Rise in threshold and exit block (Cardiac disorders) | 12 (12) | 27 (31)
Shortness of Breath (Cardiac disorders) | 11 (11) | 7 (9)
Valve damage (Cardiac disorders) | 10 (14) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 2 (3)
Diabetes (Endocrine disorders) | 12 (12) | 13 (14)
Hyperlipidemia (Endocrine disorders) | 2 (2) | 1 (1)
Hypoglycemia (Endocrine disorders) | 1 (1) | 1 (1)
Toxic multinodular goitre (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 7 (7) | 5 (7)
Galucoma (Eye disorders) | 0 (0) | 2 (2)
Macular Degeneration (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diverticulitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ulcer (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Antral gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 3 (4) | 2 (2)
Hernia (Gastrointestinal disorders) | 6 (6) | 5 (6)
Ulcerative colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Cold (General disorders) | 3 (3) | 1 (1)
Dizziness (General disorders) | 19 (19) | 13 (13)
Drug Toxicity (General disorders) | 1 (2) | 3 (3)
Dysphonia (General disorders) | 1 (1) | 0 (0)
Esophagitis (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 4 (4) | 5 (6)
Genital Prolapse (General disorders) | 1 (1) | 0 (0)
Hospitalization for non-cardiac diseases (General disorders) | 24 (26) | 18 (21)
Influenza (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 61 (87) | 53 (64)
Prolapse (General disorders) | 0 (0) | 1 (2)
Shingles (General disorders) | 3 (3) | 1 (1)
Short Loss of Consciousness (General disorders) | 0 (0) | 1 (1)
Stenosis (General disorders) | 4 (4) | 4 (4)
Syncope (General disorders) | 12 (14) | 12 (13)
Tremor (General disorders) | 1 (1) | 0 (0)
Weakness (General disorders) | 3 (3) | 1 (1)
Worsening of General Patient's Condition (General disorders) | 51 (61) | 50 (54)
Dysfibrinogenemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy (Immune system disorders) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 27 (33) | 53 (65)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Accidental injury (Injury, poisoning and procedural complications) | 4 (4) | 10 (10)
Acute hemorrhage/bleeding (Injury, poisoning and procedural complications) | 8 (9) | 15 (16)
Air emboli (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asystole during implant (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary Sinus Cannulation Failure (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cardiac or venous perforation (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Cardiac tamponade (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac/coronary sinus dissection (Injury, poisoning and procedural complications) | 0 (0) | 8 (8)
Coronary sinus or cardiac vein thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 8 (8)
Erosion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excessive bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extracardiac stimulation (phrenic nerve, diaphragm, chest wall) (Injury, poisoning and procedural complications) | 14 (14) | 77 (95)
Fall (Injury, poisoning and procedural complications) | 25 (29) | 31 (34)
Hematoma/seroma formation (Injury, poisoning and procedural complications) | 13 (13) | 29 (31)
Inverted connection of RV and LV Leads (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pericardial effusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pneumothorax (Injury, poisoning and procedural complications) | 6 (6) | 8 (8)
Steal Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Bone fracture (Musculoskeletal and connective tissue disorders) | 15 (15) | 9 (9)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gonarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7)
Hypertonia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendinitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 11 (11)
Local tissue reaction; formation of fibrotic tissue; cyst formation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 3 (3)
Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (14) | 15 (15)
Depression (Nervous system disorders) | 3 (3) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Parethesia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 3 (4) | 5 (5)
Sleep Apnea (Nervous system disorders) | 1 (2) | 0 (0)
Decreased CRT pacing (Product Issues) | 0 (0) | 1 (1)
Inability to defibrillate (Product Issues) | 0 (0) | 1 (1)
Inappropriate mode switch (Product Issues) | 1 (2) | 1 (1)
Inappropriate shocks (Product Issues) | 1 (1) | 0 (0)
Lead migration, dislodgment or poor lead placement (Product Issues) | 26 (27) | 42 (42)
Loss of Capture (Product Issues) | 6 (6) | 8 (9)
Mechanical malfunction of the pacing lead (Product Issues) | 0 (0) | 1 (1)
Oversensing (Product Issues) | 6 (7) | 6 (6)
Pacemaker Mediated Tachycardia (Product Issues) | 3 (3) | 1 (1)
Pacing Lead Impedance Out of Range (Product Issues) | 2 (2) | 4 (5)
Pulse Generator Reset (Product Issues) | 0 (0) | 2 (2)
Undersensing (Product Issues) | 5 (5) | 4 (4)
Elevated uric acid (Renal and urinary disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Prostatism (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Disease (Renal and urinary disorders) | 4 (4) | 6 (6)
Renal failure (Renal and urinary disorders) | 2 (2) | 5 (5)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Track Disease (Renal and urinary disorders) | 5 (5) | 4 (7)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 12 (12)
Nocturnal desaturation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (8)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 1 (1)
Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mastitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea on Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Colposcopy (Surgical and medical procedures) | 1 (1) | 1 (1)
Medication Titration (Surgical and medical procedures) | 0 (0) | 1 (1)
Percutaneous Coronary Intervention (Surgical and medical procedures) | 7 (7) | 9 (9)
Planned Lead Revision (Surgical and medical procedures) | 1 (1) | 0 (0)
Planned Pulse Generator Replacement (Surgical and medical procedures) | 9 (9) | 15 (15)
Pulse Generator Pocket Revision (Surgical and medical procedures) | 0 (0) | 2 (2)
Surgery (Surgical and medical procedures) | 52 (58) | 52 (64)
Aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Cerebrovascular Accident (Vascular disorders) | 3 (3) | 2 (3)
Coronary artery disease (Vascular disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Fluid accumulation (Vascular disorders) | 23 (24) | 24 (25)
Hemorrhoids (Vascular disorders) | 0 (0) | 1 (1)
Lim Ischemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2 (2) | 0 (0)
Stroke (Vascular disorders) | 3 (3) | 2 (2)
Transient Ischemic Attack (Vascular disorders) | 11 (14) | 12 (12)
Varicose Veins (Vascular disorders) | 1 (1) | 0 (0)
Venous occlusion (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less